CLINICAL TRIAL: NCT01242761
Title: Ultrasound as a Diagnostic Tool for Rotator Cuff Tears: Accuracy of Results From the Community Versus Results From a Hospital-based Ultrasound Service and Surgical Findings
Brief Title: Ultrasound as a Diagnostic Tool for Rotator Cuff Tears
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Gil Laufer, MD, Hillel Yaffe Medical Center
Other Study IDs: 0092-10-HYMC
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2010-11-17 (Estimated); Status verified 2010-11

CONDITIONS: Rotator Cuff Tear
Keywords: Accuracy of diagnostic ultrasound based in community or as part of a specialist hospital-based service
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Symptomatic rotator cuff tear: Patients with symptomatic rotator cuff tears presenting to hospital clinic after having ultrasound exam in community with indications for surgery

SUMMARY:
After comparing ultrasound study of rotator cuff injuries that have been evaluated both in the community and in a hospital-based ultrasound service with actual surgical findings, it is expected that specialist performed imaging and evaluation will be most accurate and that those performed in the community will be not accurate enough.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic rotator cuff tears Indication for rotator cuff repair

Exclusion Criteria:

* Severe arm movement limitations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptomatic rotator cuff tears
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Rotator cuff tear surgical findings more accurately reflect hospital-based US imaging findings | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel